CLINICAL TRIAL: NCT04101617
Title: Cooperation Between Dentists and Pediatricians to Improve Dental Health Among Toddlers in the Dominican Republic
Brief Title: Improving Dental Health Among Toddlers in the Dominican Republic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Iberoamericana (Other)
Collaborators: University of Copenhagen (Other); Borrow Foundation (Unknown); Hospital General Plaza de la Salud (Unknown); Colgate Palmolive (Industry)
Responsible Party: Principal Investigator, Ninoska Abreu Placeres, Researcher, Universidad Iberoamericana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEI2017-14
Record Dates: First submitted 2019-09-19; First posted 2019-09-24 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Dental Caries in Children; Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants will receive previously designed educational material with recommendations for healthy habits and oral health recommendations. Also, pediatricians will give the parents oral health education. Parents and their children will receive toothbrushes as well as toothpaste.
  Interventions: Behavioral: Oral Health education including printed educational material
- Control Group (No Intervention): Parents and their children will receive toothbrushes as well as toothpaste.

INTERVENTIONS:
Behavioral: Oral Health education including printed educational material — Printed and online educational materials were developed and provided to pediatricians so they can share relevant information about caries control to parents of toddlers. A previous interview was performed to pediatricians as focus groups to know how they are doing their evaluations and what do they take into account during the children visits in order to identify where to focus for the training what it is necessary to change. After that pediatricians were trained to give oral health recommendations. So, to the intervention group, the pediatricians will give these recommendations to the parents and also they will give them a printed educational material previously developed for the project.
  Arms: Experimental group

SUMMARY:
Caries prevalence in the Dominican Republic (DR) seems high, although recent information is lacking. In DR there is a growth and development program for all children from the age of 0 to 5.Even though there is a mandatory educational health program for children and parents in this program, where periodically pediatricians examine them, this program does not include oral health education/prevention. Thus, it is proposed A) to devise materials to be used by pediatricians to share relevant information about caries control to parents of toddlers, and B) to evaluate the impact of such material on caries prevention for groups of toddlers over a 1.5-year period. Educational material will be developed for parents, and the pediatricians will deliver this material to 10-months-old children randomly selected at Plaza de la Salud Hospital. The PI will train the pediatricians in caries prevention and how to deliver the information to the parents in a clear manner. A total of 306 will be allocated into two groups. The experimental group (128 children) will receive the devised educational materials at 10 months, follow-up information will be provided at growth and development visits when the child is 18-, and 24 months old. The second group will be considered as the control group and will not receive any educational materials (178 children). All the enrolled children will receive fluoride containing toothpaste and tooth brushes. After 18 months when the children will be about 3 years old they will be examined to assess dental caries status. A sample mortality rate of 40% is expected during the two-year follow-up. Differences in caries status between the two groups will be examined using Welch's independent t-tests for unequal variances.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children
* Parents agreed to participate in the program

Exclusion Criteria:

-

Ages: 10 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 306 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Dental caries status | Up to ten months
  Detection of dental caries lesions using the International Caries Detection and Assessment System (ICDAS) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Ekstrand, PhD, Study Director — The University of Copenhagen
Locations (1):
- Hospital General Plaza de la Salud, Santo Domingo, Nacional, Dominican Republic

IPD SHARING:
Plan to Share IPD: Undecided